CLINICAL TRIAL: NCT01551329
Title: A Randomized Controlled Trial of the N-methyl-D-aspartate (NMDA) Receptor Antagonist Ketamine in Comorbid Depression and Alcohol Dependence.
Brief Title: Ketamine for Depression and Alcohol Dependence
Acronym: KetamineDep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ismene Petrakis, Assistant Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1111009339
Record Dates: First submitted 2012-03-07; First posted 2012-03-12 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Depression; Alcohol Dependence
Keywords: depression; alcohol; comorbidity; ketamine; glutamate; NMDA
MeSH Terms: conditions — Depression; Alcoholism | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug: Ketamine (Experimental)
  Interventions: Drug: Ketalar (ketamine)

INTERVENTIONS:
Drug: Ketalar (ketamine) — Intravenous Ketamine 0.5mg/kg

SUMMARY:
The purpose of this study is to evaluate the efficacy of ketamine in reducing depressive symptoms in subjects with a comorbid major depressive episode and alcohol dependence. The investigators hypothesize the following for the present study:

A single dose of ketamine will induce a rapid, robust and sustained reduction in depressive symptoms in subjects with a comorbid major depressive episode and alcohol dependence relative to placebo as defined by change in Hamilton Depression Rating Scale total scores at 72 hours post infusion.

A single dose of ketamine can be delivered safely, with minimal adverse events or complications, in subjects with a comorbid major depressive episode and alcohol dependence.

DETAILED DESCRIPTION:
Major depression and alcohol dependence are both within the ten disorders for highest worldwide disease burden as identified by the World Health Organization (WHO), and these disorders frequently co-occur, especially in high-service utilizing patients with severe and persistent mental illness. Currently available treatments are inadequate for both chronic conditions alone, and the inadequacy is even clearer in people meeting criteria for both disorders. Ketamine was first reported as a rapidly-acting antidepressant in 2000 via research occurring at Yale, and, since that time, in several small randomized controlled trials, a single subanesthetic dose of intravenous ketamine has demonstrated efficacy in improving mood in unipolar and bipolar depression within only hours after administration. These effects can last at least a week. Interestingly, ketamine has been demonstrated to produce a more robust effect in treatment-refractory unipolar depressed subjects with a family history of alcoholism relative to similarly difficult-to-treat subjects without a family history of alcohol problems. In addition, recently-detoxified alcoholics have been safely administered subanesthetic doses of ketamine, and, during these infusions, alcoholics (and even those with only a family history of alcoholism) displayed a differential response to ketamine, e.g. blunted psychotic-like and cognitive effects, relative to healthy controls. Therefore, ketamine may reduce depressive symptoms and alcohol consumption compared to placebo in patients with comorbid major depression and current alcohol dependence. Positive results will mark a major advance in the clinical care of those being treated for both conditions and will open the door for further scientific investigations into the clinical neuroscience of these highly comorbid and prevalent conditions.

This is a two phase, double-blind, randomized, placebo-controlled, cross-over, proof-of-concept study designed to determine the effects of a single dose of ketamine, administered IV, on mood and alcohol consumption, in psychotropic medication-free patients meeting DSM-IV-TR criteria for a major depressive episode (MDE) and current alcohol dependence. Participants will be assigned randomly to receive either intravenous ketamine (0.5mg/kg) or saline solution 2 weeks apart in a cross over design. The ketamine dose was based on previous studies in patients with depression and bipolar disorder. A team member experienced with ketamine infusions will administer the study medication over a 40-minute infusion in a blinded fashion at the Biological Studies Unit at the WHVA.

20 depressed alcohol dependent subjects between the ages of 21-65 will be recruited for this study through advertising and the West Haven VA clinics. Subjects will complete an informed consent process and will be thoroughly screened for inclusion and exclusion criteria as described below. Individuals will be given a post consent test to evaluate their understanding of the procedure. For subjects who provide incorrect answers to any of the test items, the research staff will review the correct answers with the subject and show the subject where the correct answers are found in the consent form. Those who get more than 60% of the questions wrong and are still unable to understand the procedure after reviewing it with the research staff will be excluded from the study. They will be referred to appropriate resources for outpatient treatment of their depression and alcoholism. Before start of the study all patients will be free of any psychotropic medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (post-menopausal, surgically sterile or negative pregnancy test at screening and agreement to utilize a medically-approved birth control method including complete abstinence during the testing period) between the age of 21 and 65 years old.
2. Able to provide written informed consent according to the WHVA and Yale HIC guidelines.
3. Medically and neurologically healthy on the basis of medical history, physical examination, EKG, and screening laboratories (CBC w/ differential, basic metabolic profile including BUN/creatinine, TSH, fT4, AST, ALT, GGT, total protein, albumin, vitamin B12, folate, VDRL, HIV, hepatitis B and C, urinalysis, HCG, and urine toxicology screen). Predefined exclusion criteria are identified, e.g. LFTs > 3x upper limit of normal. Individuals with stable medical problems that do not have direct CNS effects, e.g. hypertension and diabetes mellitus, or interfere with medications administered, e.g. oral hypoglycemics, may be included if their medications have not been adjusted in the month prior to study enrollment.
4. Current DSM-IV-TR major depressive episode (MDE) by structured clinical interview (SCID) and a MADRS score ¬>20.
5. Current DSM-IV-TR alcohol dependence with one heavy drinking day (> 4 standard drinks/session for men and > 3 standard drinks/session for women) in the last 3 weeks.
6. Abstinent from drinking for > 5 days prior to receiving ketamine.
7. No current psychotropic medications (excluding benzodiazepines during alcohol detoxification if needed) in last 2 weeks (4 weeks for fluoxetine).
8. Individuals who have completed a detoxification program and who are at least 5 days past their last drink.

Exclusion Criteria:

1. Unstable medical condition or medical problem with known CNS effects, e.g. uncontrolled hypertension (SBP≥170 and/or DBP≥100) or confirmed history of alcohol-withdrawal seizures.
2. Active suicidal ideation, intent or plan.
3. Active DSM-IV-TR substance use disorder in past three months (other than an alcohol or nicotine use disorder).
4. Prior diagnosis of a DSM-IV-TR psychotic spectrum disorder, e.g. schizophrenia, schizoaffective disorder, bipolar I d/o with psychotic features, MDD with psychotic features.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Depression | 29 Days
  Measured using the Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA CT Healthcare Systems, West Haven, Connecticut, United States